CLINICAL TRIAL: NCT04368598
Title: The Combination of High-dose Dexamethasone and Acetylcysteine as the Treatment of Newly-diagnosed Immune Thrombocytopenia: A Single-arm, Open-label Trial
Brief Title: The Combination of High-dose Dexamethasone and Acetylcysteine as the Treatment of Newly-diagnosed ITP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITP-PKU008
Record Dates: First submitted 2020-04-26; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Immune Thrombocytopenia
Keywords: immune thrombocytopenia; acetylcysteine
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone; Acetylcysteine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-dose Dexamethasone plus Acetylcysteine (Experimental): For all patients in this arm, DXM was administered intravenously at 40 mg daily for 4 consecutive days and then stopped. If platelet count remained below 30×10^9/L or there were bleeding symptoms by day 10 to 14, an additional 4-day course of DXM (40 mg daily) was given. Besides, all patients received Acetylcysteine orally at 0.4g three times a day for 4 consecutive weeks in the first month.
  Interventions: Drug: Dexamethasone; Drug: Acetylcysteine

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone, iv, 40 mg/d, for 4 days (The 4-day course of dexamethasone was repeated on days 11 to 14 in the case of lack of response by day 10)
  Other Names: HD-DXM; High-dose Dexamethasone
Drug: Acetylcysteine — Acetylcysteine, po, 400mg tid, for 4 weeks
  Other Names: YiWeiShi

SUMMARY:
A single-arm, open-label study to evaluate the efficacy and safety of Acetylcysteine plus high-dose Dexamethasone in adults newly diagnosed with primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
This is a prospective, open-label, Phase II, single-arm interventional trial performed in a single center in China. The investigators explore the efficacy and safety of Acetylcysteine plus high-dose Dexamethasone in adults newly diagnosed with primary immune thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically confirmed immune thrombocytopenic purpura (ITP) newly diagnosed
2. Platelet count less than 30×10^9/L on two occasions or Platelets above 30×10^9/L combined with bleeding manifestation (WHO bleeding scale 2 or above)
3. Subject is ≥ 18 years and ≤80years
4. Subject has signed and dated written informed consent.
5. Fertile patients must use effective contraception during treatment and observational period
6. Negative pregnancy test

Exclusion Criteria:

1. Have an impaired renal function as indicated by a serum creatinine level > 2.0 mg/dL
2. Have an inadequate liver function as indicated by a total bilirubin level > 2.0 mg/dL and/or an aspartate aminotransaminase or alanine aminotransferase level > 3×upper limit of normal
3. Have a New York Heart Classification III or IV heart disease
4. Have a history of severe psychiatric disorder or are unable to comply with study and follow-up procedures
5. Have active hepatitis B or hepatitis C infection
6. Have a HIV infection
7. Have active infection requiring antibiotic therapy within 7 days prior to study entry
8. Are pregnant or lactating women, or plan to become pregnant or impregnated within 12 months of receiving study drug
9. Previous treatment with rituximab
10. Previous splenectomy
11. Had previous or concomitant malignant disease
12. Not willing to participate in the study.
13. Expected survival of < 2 years
14. Intolerant to murine antibodies
15. Immunosuppressive treatment within the last month
16. Connective tissue disease
17. Autoimmune hemolytic anemia
18. Patients currently involved in another clinical trial with evaluation of drug treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with durable response after 6 months | 6 months
  Number of patients with durable response after 6 months

SECONDARY OUTCOMES:
Early response | 7 days
  Number of patients with early response on day 7
Initial response | 1 month
  Number of patients with initial response at 1 month
Bleeding | 1 year
  Number of patients with bleeding complication therapy; bleeding score
DOR | 1 year
  duration of response
Relapse | 1 year
  Number of patients relapse during the observation
Adverse events | 1 year
  Number of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, MD, Principal Investigator — Peking University People's Hospital, Peking University Insititute of Hematology
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No